CLINICAL TRIAL: NCT05948852
Title: Randomized Prospective Study Comparing Two Hypoabsorption Techniques for the Treatment of Type III Obesity (Body Mass Index Between 45 - 49.9 Kg/m2): Single Anastomose Duodenal Switch (SADI-S) and Single Anastomose Gastric By-pass (OAGBP)
Brief Title: Two Hypoabsorption Techniques for the Treatment of Type III Obesity (OASIS)
Acronym: OASIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23/001
Record Dates: First submitted 2023-06-12; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Obesity, Morbid
Keywords: OAGB; SADIS; bariatric surgery
MeSH Terms: conditions — Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: SADI-S (Experimental): SINGLE ANASTOMOSE DUODENAL SWITCH
  Interventions: Procedure: metabolic surgery (SADIS and OAGB)
- Group B: OAGB (Active Comparator): SINGLE ANASTOMOSE GASTRIC BY-PASS
  Interventions: Procedure: metabolic surgery (SADIS and OAGB)

INTERVENTIONS:
Procedure: metabolic surgery (SADIS and OAGB) — TWO HYPOABSORPTION TECHNIQUES FOR THE TREATMENT OF TYPE III OBESITY (BODY MASS INDEX BETWEEN 45 - 49.9 KG/M2): SINGLE ANASTOMOSE DUODENAL SWITCH (SADI-S) AND SINGLE ANASTOMOSE GASTRIC BY-PASS (OAGBP).

SUMMARY:
This study aims to compare the percentage of total weight lost in long-term follow-up after two surgical interventions (SADIS and OAGB) in patients with morbid obesity BMI between 45-49.9.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 and under 65 who meet criteria for bariatric surgery.
* Maximum BMI between 45 and 50 kg/m2 and indication for surgery in a time
* Signature of the informed consent of the study
* Patients suitable for laparoscopic surgery

Exclusion Criteria:

* Previous bariatric surgery
* 2-stage surgery
* Contraindication for hypoabsorptive surgery due to previous pathology: inflammatory bowel disease, transplant recipient or transplant candidate, previous intestinal resection surgery
* Other associated surgical procedures in the same intervention.
* Conversion to laparotomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
the percentage of total weight loss (%TWL) of the patients after surgery | Baseline, 1 year, 3 year, 5 year after SADI-S and OAGBP surgery

SECONDARY OUTCOMES:
% of patients with gastroesophageal reflux (acid and bile) after surgery | 1 year, 3 year, 5 year after SADI-S and OAGBP surgery
Number of deaths in the immediate postoperative period | up to day 90 post-intervention
Number of Participants with complications in the immediate postoperative period | up to day 90 post-intervention
Ratio of patients with more than 3 loose stools per day | 1 year, 3 years, 5 years after the surgery
  The ratio of patients with more than 3 loose stools per day will be evaluated as pathological. To assess the quality of the bowel movements, the Bristol Stool Form Scale questionnaire will be used. An evaluation of the number of bowel movements and their quality according to the Bristol Stool Form Scale questionnaire will be conducted at 1 year, 3 years, and 5 years after the surgery
questionnaire of quality of life | 1 year, 3 years, 5 years after SADI-S and OAGBP surgery
  The quality of life will be assessed based on the results of the Moorehead-Ardelt II test and the Medical Outcomes Study Short Form-36 questionnaire. The Moorehead-Ardelt II questionnaire includes 6 parameters related to self-esteem, physical activity, social contact, job satisfaction, sexual pleasure, and eating habits. The minimum score is -3 and the maximum is +3. A score of 1.1 to 2 is considered a good result, and anything above 2.1 is considered very good.
  The SF-36 questionnaire includes 8 parameters such as physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The minimum score is 0 and the maximum is 100.
Number of patients with nutritional deficiencies | 1 year, 3 years, 5 years after SADI-S and OAGBP surgery
  The main nutritional deficiencies to be evaluated after OAGB (One Anastomosis Gastric Bypass) and SADIS (Single Anastomosis Duodeno-Ileal Switch) are iron and/or vitamin B12 deficiency anemia, deficiencies in fat-soluble vitamins, calcium, and trace elements.
  The incidence of nutritional deficiencies will be assessed through routine blood tests at 1 year, 3 years, and 5 years after the surgery

IPD SHARING:
Plan to Share IPD: No